CLINICAL TRIAL: NCT06992076
Title: Adult and Adolescent Hemophilia Patients Treated With Marstacimab: a Patient Experience Registry
Acronym: AMBER
Status: Not yet recruiting | Type: Observational
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Other Study IDs: QT2025001
Record Dates: First submitted 2025-05-19; First posted 2025-05-28 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-05

CONDITIONS: Hemophilia
MeSH Terms: conditions — Hemophilia A | interventions — marstacimab

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Marstacimab — the first visit (V1) is scheduled on the day of the first administration of marstacimab. The recommended dosing frequency for the patient should follow the instructions provided, which are as follows: On Day 1, administer 300 mg subcutaneously (divided into two injections, each 150 mg) (loading dose); starting from Day 8, administer 150 mg subcutaneously once a week. Record the patient's prescription recommendations, actual treatment records (administration time, dosage, frequency), and adherence rates. Visit 2 (V2) and visit 3 (V3) are defined as 30 days (±7 days) and 180 days (±30 days) after the initiation of marstacimab treatment, respectively.

SUMMARY:
Research Title：Adult and adolescent hemophilia patients treated with Marstacimab: a patient Experience Registry (AMBER) Protocol Number：94250855 Protocol Version Number：version 0.3 Date：15-November-2024 Leading site：Institution of Hematology & Blood Diseases Hospital, Chinese Academy of Medical Sciences Active Pharmaceutical Ingredient：a human IgG1 monoclonal antibody that targets the tissue factor pathway inhibitor (TFPI) Drug Name Generic name: marstacimab-hncq Purpose of the Study Primary Objectives:To quantify patient preferences for subcutaneous versus intravenous (IV) injection using the Marstacimab-Patient Preference Questionnaire (M-PPQ) after 1 month of marstacimab for routine prophylaxis treatment.

To assess the treatment burden using the Hemophilia Treatment Experience Measure (Hemo-TEM) in hemophilia patients after 6 months of marstacimab for routine prophylaxis treatment.

Exploratory Objectives:

To evaluate the annualized bleeding rate (ABR) of different types of bleeds after 6 months of subcutaneous marstacimab injections in hemophilia patients.

To assess changes in joint status scores between baseline and the final visit after 6 months of subcutaneous marstacimab injections in hemophilia patients, using the Hemophilia Early Arthropathy Detection with Ultrasound in China (HEAD-US-C).

To evaluate patient preferences regarding treatment experience via M-PPQ after 6 months

ELIGIBILITY:
Inclusion Criteria:

- Participants with a diagnosis of hemophilia A or hemophilia B eligible to receive prophylaxis.

Clinical physicians prescribe marstacimab for routine prophylaxis treatment of hemophilia patients based on the actual conditions of the patients and in accordance with the approved indications of marstacimab.

Adolescent patients(12 to less than 18 years) and adult (18 years and older) patients.

Signed consent obtained before the study, participant or legally authorized representative, or participant's caregiver capable of giving signed informed consent.

Exclusion Criteria:

- Those who are unable to complete at least one month follow-up based on the investigator's judgment.

Severe impairment of speech, vision, memory or cognition that affects communication and ability to complete questionnaires and follow-up visits.

Women of childbearing age who plan to become pregnant within the next 2 months, as well as women who are pregnant or breastfeeding.

Patients are participating in other clinical trials. There are other conditions that the investigator deems unsuitable for participation in this study.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with hemophilia who will receive marstacimab for routine prophylactic treatment in a real-world setting. Each patient will receive treatment and care according to the standard clinical practice. The total recruitment period will be 18 months. Patients will be prescribed marstacimab in routine practice and initiate marstacimab treatment on the same day (or as soon as possible after prescribing). The observation period for individual patients is defined as ending on the 180th day from the index date (the date of the first dose of marstacimab).
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-08-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
patient preferences for subcutaneous | after 1 month of marstacimab treatment
  To quantify patient preferences for subcutaneous versus intravenous (IV) injection using the Marstacimab-Patient Preference Questionnaire (M-PPQ) after 1 month of marstacimab for routine prophylaxis treatment.
To assess the treatment burden | after 6 month of marstacimab treatment
  To assess the treatment burden using the Hemophilia Treatment Experience Measure (Hemo-TEM) in hemophilia patients after 6 months of marstacimab for routine prophylaxis treatment.

SECONDARY OUTCOMES:
To evaluate the annualized bleeding rate (ABR) | after 6 month of marstacimab treatment
  To evaluate the annualized bleeding rate (ABR) of different types of bleeds after 6 months of subcutaneous marstacimab injections in hemophilia patients.
To assess changes in joint status scores | after 6 month of marstacimab treatment
  To assess changes in joint status scores between baseline and the final visit after 6 months of subcutaneous marstacimab injections in hemophilia patients, using the Hemophilia Early Arthropathy Detection with Ultrasound in China(HEAD-US-C).
patient preferences for subcutaneous | after 6 month of marstacimab treatment
  To evaluate patient preferences regarding treatment experience via M-PPQ after 6 months.

IPD SHARING:
Plan to Share IPD: No
Patient-level variables including demographics, clinical characteristics, treatment history will be extracted from medical records. Patient-reported outcomes (PROs), namely the M-PPQ and Hemo-TEM questionnaires, will be reported by patients. Clinician-reported outcomes (ClinROs), namely the HEAD-US-C scale, will be reported by clinicians who have undergone training and certification. Electronic case report forms (eCRFs) will be prepared for all data collection fields.